CLINICAL TRIAL: NCT02618174
Title: Enhanced Broccoli Consumption After a Liking Norm and Vegetable Variety Message: Effects After a 24 Hour Delay.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UBirmingham-SNS1
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Eating Behaviour
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Neutral Control Condition (Placebo Comparator): Message about age of University of Birmingham
  Interventions: Behavioral: Neutral Control Condition
- Food-based Control Condition (Placebo Comparator): Message about variety of vegetables in the world
  Interventions: Behavioral: Food-based Control Condition
- Health Condition (Active Comparator): Message about the health benefits of eating vegetables
  Interventions: Behavioral: Health Condition
- Descriptive Social Norm (Active Comparator): Message suggesting most people eat plenty of vegetables
  Interventions: Behavioral: Descriptive Social Norm
- Liking Social Norm (Experimental): Message suggesting most people like eating vegetables
  Interventions: Behavioral: Liking Social Norm

INTERVENTIONS:
Behavioral: Neutral Control Condition — Message about age of University of Birmingham
  Arms: Neutral Control Condition
Behavioral: Food-based Control Condition — Message about variety of vegetables in the world
  Arms: Food-based Control Condition
Behavioral: Health Condition — Message about the health benefits of eating vegetables
  Arms: Health Condition
Behavioral: Descriptive Social Norm — Message suggesting most people eat plenty of vegetables
  Arms: Descriptive Social Norm
Behavioral: Liking Social Norm — Message suggesting most people like eating vegetables
  Arms: Liking Social Norm

SUMMARY:
Encouraging individuals to eat vegetables is difficult. However, recent evidence suggests that using social-based information might help. For instance, it has been shown that if people think that others are eating lots of fruit and vegetables, that they will consume more of these foods to match the 'norm'. The purpose of this study was to determine whether a liking social norm (information about how much others like vegetables) would be effective at encouraging people to eat more vegetables and to examine whether these effects are sustained beyond initial exposure (i.e. whether the effect of the norm persists on food selection 24 hours alter).

DETAILED DESCRIPTION:
Using a 2 x 5 x 2 experimental design we investigated the effects of exposure to various messages on later food intake and whether any effects were sustained 24 hours after exposure in both low and high consumers of vegetables. There were three factors of delay (immediate food selection versus food selection 24 hours after exposure), message type (liking norm, descriptive norm, health message, food-based control, and neutral control message) and habitual consumption (low versus high). The buffet consisted of three raw vegetables, three energy-dense foods and two dips.

In this study the investigators hypothesised that a liking norm would increase the consumption of vegetables (compared to a neutral control condition) and that the effect would persist on vegetable consumption 24 hours after intital exposure to the liking norm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Sufficiently fluent in English

Exclusion Criteria:

* Smokers
* Diabetes
* Food allergies
* Past / present depression or anxiety
* Past / present eating disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Grams of vegetables consumed | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Thomas, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Thomas JM, Liu J, Robinson EL, Aveyard P, Herman CP, Higgs S. The Effects of Liking Norms and Descriptive Norms on Vegetable Consumption: A Randomized Experiment. Front Psychol. 2016 Mar 30;7:442. doi: 10.3389/fpsyg.2016.00442. eCollection 2016. PMID 27065913